CLINICAL TRIAL: NCT05600283
Title: Validation and Feasibility of Patient Self-sampling of HPV for Cervical Cancer Screening
Brief Title: Patient Self-sampling of HPV to Screen for Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 22-008247; NCI-2022-10804 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2024-10

CONDITIONS: Human Papilloma Virus
Keywords: Cervical Cancer Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self-collected vaginal swab samples (Experimental): Subjects will self-collect a vaginal swab (Evalyn brush) and complete a scheduled standard of care clinician-collected cervical swab
  Interventions: Diagnostic Test: Swab kit (COBAS HPV 4800 Assay -Evalyn brush); Diagnostic Test: Clinician-collection of cervical sample for HPV testing

INTERVENTIONS:
Diagnostic Test: Swab kit (COBAS HPV 4800 Assay -Evalyn brush) — Patient self-sampling swab kit to collect a vaginal sample for HPV testing
Diagnostic Test: Clinician-collection of cervical sample for HPV testing — Speculum exam and collection of a cervical specimen using standard endocervical brush and spatula placed into ThinPrep medium for HPV testing (Evalyn brush)

SUMMARY:
The purpose of this study is to validate a patient self-sampling vaginal collection kit and laboratory testing for the detection of HPV (human papillomavirus) infection. Researchers will compare the laboratory results of self-collected vaginal swab samples to usual healthcare provider-collected cervical swab samples to determine the laboratory HPV testing accuracy of the self-collection swab.

ELIGIBILITY:
Inclusion Criteria:

* Appointment at Mayo Clinic Rochester in Gynecology Colposcopy Clinic or ICS (integrated community specialty) Colposcopy Clinic (will always include a speculum exam).
* Appointment at Mayo Clinic Rochester in Gynecology Clinic for indication that will already include a speculum exam (e.g., cervical cancer screening or IUD insertion).

Exclusion Criteria:

* Excluded if self-reported as currently menstruating, pregnant, or within 3 months following pregnancy.
* Excluded if no cervix (history of total hysterectomy).
* Excluded if moderate to heavy vaginal bleeding on the day of the visit.
* Excluded if reason for visit in Gynecology Clinic is abnormal vaginal discharge.
* Exclude patients who are on Gynecology Colposcopy Clinic for LEEP (loop electrosurgical excision procedure).
* Exclude if any use of over-the-counter or prescription vaginal cream for vaginal infection or prescription vaginal estrogen cream for at least two days before using the Evalyn Brush.

(Vaginal contraceptives, condoms and water-based lubricants can be used as normal.)

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy MacLaughlin, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Group 1: eligible participants enrolled = 89 (98 participants initially deemed eligible; 9 participants declined to participate) Group 2: eligible participants enrolled = 133 (207 participants initially deemed eligible; 74 declined to participate)
Groups:
- Group 1: Self-collected Vaginal Swab Samples at Clinic; Group 2: Self-collected Vaginal Swab Samples at Home: Subjects will self-collect a vaginal swab (Evalyn brush) and complete a scheduled standard of care clinician-collected cervical swab
  Swab kit (COBAS HPV 4800 Assay -Evalyn brush): Patient self-sampling swab kit to collect a vaginal sample for HPV testing
  Clinician-collection of cervical sample for HPV testing: Speculum exam and collection of a cervical specimen using standard endocervical brush and spatula placed into ThinPrep medium for HPV testing (Evalyn brush)
Period: Overall Study
Arm/Group | Group 1: Self-collected Vaginal Swab Samples at Clinic | Group 2: Self-collected Vaginal Swab Samples at Home
Started | 89 | 133
Completed | 79 | 115
Not Completed | 10 | 18
Not completed — Withdrawal by Subject | 3 | 8
Not completed — Invalid Vaginal Swab | 2 | 2
Not completed — Missing Clinician Collection | 3 | 6
Not completed — Screen Failure | 1 | 2
Not completed — Sample Lost in Transit | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Self-collected Vaginal Swab Samples at Clinic | Group 2: Self-collected Vaginal Swab Samples at Home | Total
Number analyzed (Participants) | 81 | 127 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 81 | 127 | 208
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 127 | 208
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 77 | 122 | 199
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 3 | 3
  White | 72 | 114 | 186
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 81 | 127 | 0

OUTCOME MEASURES:

1. Primary Outcome: Concordance of Patient-collected and Clinician-collected Samples to Detect HPV Infection
Description: Patient-collected vaginal swab HPV results compared with gold standard of clinician-collected cervical swab) to accurately detect HPV infection
Time Frame: Baseline (sample was collected up to 21 days form the date of registration)
Measure: Number; unit: Total Percentage Agreement
Arm/Group | Group 1: Self-collected Vaginal Swab Samples at Clinic | Group 2: Self-collected Vaginal Swab Samples at Home
Number analyzed (Participants) | 79 | 115
Total Percentage Agreement
  HPV16 | 98 | 94
  HPV18 | 99 | 95
  Other HPV | 86 | 89

2. Secondary Outcome: Patient-reported Acceptability of Using the Evalyn Brush
Description: Assessed by survey question "Overall, how acceptable was it for you to collect the sample using the Evalyn® brush?," which was answered on a 4-point scale (completely unacceptable, unacceptable, acceptable, or completely acceptable).
Time Frame: Baseline (sample was collected up to 21 days form the date of registration)
Population: Survey results are reported for all participants who completed vaginal self-collection and returned the survey, even if the self-collection sample was deemed invalid or clinician sample was not received.
Measure: Number; unit: Participants
Arm/Group | Group 1: Self-collected Vaginal Swab Samples at Clinic | Group 2: Self-collected Vaginal Swab Samples at Home
Number analyzed (Participants) | 81 | 126
Participants
  Completely unacceptable | 0 | 0
  Unacceptable | 0 | 1
  Acceptable | 15 | 37
  Completely acceptable | 66 | 88

ADVERSE EVENTS:
Time Frame: Baseline (at the time of swab collection). Participants collected swab samples up to 21 days from the time of enrollment.
Arm/Group | Group 1: Self-collected Vaginal Swab Samples at Clinic | Group 2: Self-collected Vaginal Swab Samples at Home
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/127
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/127
Other Adverse Events (participants affected / at risk) | 2/81 | 1/127
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Self-collected Vaginal Swab Samples at Clinic (N=81) | Group 2: Self-collected Vaginal Swab Samples at Home (N=127)
Participant inserted self-collection device with cap on (did not remove cap) (Product Issues) | 2 (2) | 0 (0) — No harm resulted from events. The study team thereafter highlighted the instruction sheet where it tells the subject to remove the cap.
Device damaged during mailing to patient (Product Issues) | 0 (0) | 1 (1) — Participant unable to rotate vaginal brush, even with additional pressure. Device broke as it was withdrawn. Manufacturer verified no defect with product at shipment. Following event, devices were mailed in boxes instead of padded envelopes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT05600283/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT05600283/ICF_001.pdf